CLINICAL TRIAL: NCT03790527
Title: A Research on the Mechanism of Cognitive Bias Modification Training in Internet Gaming Disorders.
Brief Title: Cognitive Bias Modification Training on Internet Gaming Disorder
Acronym: CBM&IGD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, Jin-tao Zhang, Associated Professor, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IGD_CBM intervention
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: The investigators assigned subjects to two training groups and collected pre - and post-test data
Who Masked: Participant, Investigator
Masking Description: double blind: both participants and experimenters won't know which group is training group or sham control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBM training (Experimental): participants have to complete the picture assessment task ; Approach-avoidance Task(AAT) and cue-induced task in the fMRI；data on game-craving level, game hours, the ability of self-control and emotion regulation are also collected.
  Half of the participants will be random-assigned into the CBM training group; Each participant will do these task twice( e.g. Before training and after training)
  Interventions: Procedure: CBM training
- Sham training (Sham Comparator): participants have to complete the picture assessment task ; Approach-avoidance Task(AAT) and cue-induced task in the fMRI；data on game-craving level, game hours, the ability of self-control and emotion regulation are also collected.
  Half of the participants will be random-assigned into the sham training group; Each participant will do these task twice( e.g. Before training and after training)
  Interventions: Procedure: Sham training

INTERVENTIONS:
Procedure: CBM training — participants will be random-assigned into one of training groups. Participants in the modification group will receive modified training of 400 trials for six sessions during six days, the same as the sham group.The difference between these two groups is the proportion of push/pull trials. The sequence of the interventions will be counterbalanced across participants, and the callback will be conduct after one week.
  Arms: CBM training
Procedure: Sham training — participants will be random-assigned into one of training groups. Participants in the modification group will receive modified training of 400 trials for six sessions during six days, the same as the sham group.The difference between these two groups is the proportion of push/pull trials. The sequence of the interventions will be counterbalanced across participants, and the callback will be conduct after one week.
  Arms: Sham training

SUMMARY:
To investigate whether and how the CBM training will alleviate the symptoms of addiction in Internet gaming disorders.

DETAILED DESCRIPTION:
The purpose of this study is to use the modification training of cognitive bias to ameliorate the severity and symptoms of Internet gaming disorders(IGD); the neural mechanisms of cognitive bias modification and its effect during cued-induced craving task in subjects with IGD will be investigated as well. This project will be conducted in Beijing, China.

ELIGIBILITY:
Inclusion Criteria:

1, DSM-5 recommended diagnosis of Internet gaming disorder :

1. the scores of the 9 items of DSM-5 recommended diagnosis for Internet gaming disorder ≥ 5.
2. engagement in popular Internet games (e.g. Arena of Valor, League of Legends and Player Unknown's Battle Grounds) for over 20 hours per week for a minimum of 12 months.

2, the scores of the Y-IAT(Young-Internet addiction Test) ≥ 50

Exclusion Criteria:

current or history of use of illegal substances and gambling;

current or history of psychiatric or neurological illness;

current use of psychotropic medications.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-13 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral outcome | 60- 80 minutes after training
  Cognitive bias outside fMRI measured by AAT task takes the response times[[Push_game_pic-Pull_game_pic]-[Push_object_pic - Pull_object_pic])] as the index. The response times (cognitive bias scores) will be calculated under Repeated Measurement Anova by using SPSS software.
Resting-state functional connectivity alterations in brain. | 30-45 minutes after training
  Using seed-based and network level functional connectivity analysis, as well as graph theory analysis , functional connectivity in brain under eight minutes resting state will be detected and compared between CBM training group and sham group
task-based fMRI brain activation | 45-60 minutes after training
  The active of the brain regions in mPFC and VS during AAT task changes after CBM training compared with the sham. There should be an decrease in ventral striatum and amygdala during the cue-induced task. These task-based fMRI data will be contrasted using SPM.
Correlation analysis | 30- 60 minutes after training
  The correlation between functional network organization in brain across resting state ( task-based fMRI) and cognitive bias scores will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tao Zhang, PhD, Principal Investigator — Beijing Normal University
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wiers CE, Stelzel C, Gladwin TE, Park SQ, Pawelczack S, Gawron CK, Stuke H, Heinz A, Wiers RW, Rinck M, Lindenmeyer J, Walter H, Bermpohl F. Effects of cognitive bias modification training on neural alcohol cue reactivity in alcohol dependence. Am J Psychiatry. 2015 Apr;172(4):335-43. doi: 10.1176/appi.ajp.2014.13111495. Epub 2014 Dec 19. PMID 25526597
- [Background] Wiers CE, Ludwig VU, Gladwin TE, Park SQ, Heinz A, Wiers RW, Rinck M, Lindenmeyer J, Walter H, Bermpohl F. Effects of cognitive bias modification training on neural signatures of alcohol approach tendencies in male alcohol-dependent patients. Addict Biol. 2015 Sep;20(5):990-9. doi: 10.1111/adb.12221. Epub 2015 Jan 13. PMID 25639749
- [Background] Rinck M, Becker ES. Approach and avoidance in fear of spiders. J Behav Ther Exp Psychiatry. 2007 Jun;38(2):105-20. doi: 10.1016/j.jbtep.2006.10.001. Epub 2006 Nov 28. PMID 17126289